CLINICAL TRIAL: NCT06898424
Title: Effects of Concurrent Plant-Based Ketogenic Diet and Intermittent Fasting (Ketoflex 12/3) on the Clinical Progression of Early-to-Mid Stage Alzheimer's Dementia
Brief Title: Impact of Ketoflex 12/3 Diet on Early-to-Mid Stage Alzheimer's Progression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Lutfu Hanoglu, MD (Other)
Responsible Party: Sponsor-Investigator, Prof. Lutfu Hanoglu, MD, Prof. MD, Istanbul Medipol University Hospital
Organization: Istanbul Medipol University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ALZ23992
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Type Dementia; Alzheimer's Disease (AD)
Keywords: Alzheimer's Disease; Ketogenic Diet; Intermittent Fasting; Ketoflex 12/3; Cognitive Decline; Neurodegeneration
MeSH Terms: conditions — Alzheimer Disease; Intermittent Fasting; Cognitive Dysfunction; Nerve Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketoflex 12/3 Diet Group (Experimental): Participants follow the Ketoflex 12/3 dietary protocol.
  Interventions: Behavioral: Ketoflex 12/3 Diet
- Control Group (No Intervention): Participants continue their usual diet with no modifications

INTERVENTIONS:
Behavioral: Ketoflex 12/3 Diet — plant-based ketogenic diet combined with intermittent fasting (12/3)
  Arms: Ketoflex 12/3 Diet Group

SUMMARY:
This study investigates the effects of the Ketoflex 12/3 diet on the clinical progression of early-to-mid stage Alzheimer's disease. The study evaluates cognitive function, metabolic changes, and overall health outcomes in participants following the Ketoflex 12/3 dietary protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50-85 years
* Clinical Dementia Rating (CDR) score of 0.5 or 1
* Diagnosis of Alzheimer's disease (AD) according to NINCDS-ADRDA criteria

Exclusion Criteria:

* Alcohol and/or substance dependence
* Diagnosis of chronic renal failure
* Diagnosis of another neuropsychiatric disorder
* Presence of amalgam dental fillings and/or failure to have them removed following the SMART protocol

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive Function as Measured by the MMSE Score | Baseline and 6 months
  Mini-Mental State Examination (MMSE) will be used to assess cognitive function before and after the intervention.
  The Mini-Mental State Examination (MMSE) is used to assess cognitive function. The total score ranges from 0 to 30, with higher scores indicating better cognitive performance.

CONTACTS AND LOCATIONS:
Overall Officials: Lütfü Hanoğlu, Prof. MD, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol Universitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
At this time, no final decision has been made regarding individual participant data (IPD) sharing. Future data-sharing plans will be considered in accordance with institutional policies, ethical guidelines, and publication requirements